CLINICAL TRIAL: NCT03556631
Title: Effect of Live Combined Bifidobacterium and Lactobacillus on Glycemic Control and Other Diabetes-Related Outcomes in People With Type 1 Diabetes:a Single-blind Randomized Controlled Trial
Brief Title: Effect of Live Combined Bifidobacterium and Lactobacillus on Glycemic Control and Other Outcomes in Type 1 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SZLY2018009
Record Dates: First submitted 2018-05-22; First posted 2018-06-14 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Type 1 Diabetes Mellitus; Probiotics
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Lacteol; Probiotics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- probiotics group (Experimental): live combined Bifidobacterium and Lactobacillus tablets were given to the participants according to their group assignment ,4 tablets ,tid, for 3 months
  Interventions: Drug: live combined Bifidobacterium and Lactobacillus Tablets
- placebo group (Placebo Comparator): placebo were given to the participants according to their group assignment ,4 tablets ,tid, for 3 months
  Interventions: Drug: live combined Bifidobacterium and Lactobacillus Tablets

INTERVENTIONS:
Drug: live combined Bifidobacterium and Lactobacillus Tablets — take the live combined Bifidobacterium and Lactobacillus Tablets 4# or placebo twice a day
  Other Names: probiotics

SUMMARY:
Aim Evidence of a possible connection between gut microbiota and several physiological processes linked to type 1 diabetes is increasing. However, the effect of multistrain probiotics in people with type 1 diabetes remains unclear. This study investigated the effect of live combined Bifidobacterium and Lactobacillus preparation on glycemic control and other diabetes-related outcomes in people with type 1 diabetes.

DETAILED DESCRIPTION:
Design A randomized, single-blind, parallel-group, controlled clinical trial. Setting Diabetes clinic of a teaching hospital in Shenzhen China Participants A total of 30 participants with type 1 diabetes, aged 18-60 years, will be recruited and randomly assigned to receive either probiotics (n = 15) or placebo (n = 15) for 12 weeks.

Outcomes Primary outcomes were glycemic control related parameters, and secondary outcomes were anthropomorphic variables, lipid profile, blood pressure and high-sensitivity C-reactive protein. The gut microbiota profile will be analyzed before and after intervention and between groups.

ELIGIBILITY:
Inclusion Criteria:

type 1 diabetes patients ,age 18-60years old,18 Kg/m2≤BMI≤30Kg/m2, 7.0mmol/L<fasting blood glucose <13.0mmol/L；HbA1c≤10%，ketonuria (-)；

Exclusion Criteria:

pregnancy, lactation, having other severe chronic illnesses.taking other anti-diabetic drugs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
hemoglobin A1c in percentage | 3 months
  analyze the change of hemoglobin A1c between two groups

SECONDARY OUTCOMES:
weight in kilograms | 3 months
  analyze the change of weight in kilograms between two groups

CONTACTS AND LOCATIONS:
Overall Officials: Ping Xu, Principal Investigator — associate chief physician
Locations (1):
- Shenzhen People' S Hospital, Shenzhen, China

IPD SHARING:
Plan to Share IPD: Undecided